CLINICAL TRIAL: NCT06784726
Title: Odronextamab for Relapsed/Refractory Large B-cell Lymphomas Before Definitive Lymphoma-Directed Therapies
Brief Title: Odronextamab for Relapsed and Refractory Large B-cell Lymphomas Before CAR-T
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1124641; NCI-2024-10534 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020747 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Recurrent Grade 3b Follicular Lymphoma; Recurrent High Grade B-Cell Lymphoma; Recurrent Primary Mediastinal Large B-Cell Lymphoma; Recurrent Transformed Indolent B-Cell Non-Hodgkin Lymphoma to Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Refractory Grade 3b Follicular Lymphoma; Refractory High Grade B-Cell Lymphoma; Refractory Primary Mediastinal Large B-Cell Lymphoma; Refractory Transformed Indolent B-Cell Non-Hodgkin Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Specimen Handling; Biopsy; Immunotherapy, Adoptive; Leukapheresis; Spinal Puncture; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (odronextamab) (Experimental): Patients receive odronextamab IV based on the following schedules:
  * Step-up dosing during cycle 1: 0.2 mg on C1D1, 0.5 mg on C1D2, 2 mg on C1D8 and C1D9, respectively, and 10 mg on C1D15 and C1D16, respectively (0.7/4/20 regimen).
  * Dosing during cycles 2-4: Odron will be given at 160 mg weekly.
  * Once every other week at 320 mg of remaining cycles.
  Please see the Detailed Description for additional information.
  Interventions: Biological: Odronextamab; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Biological: Chimeric Antigen Receptor T-Cell Therapy; Procedure: Computed Tomography; Procedure: Leukapheresis; Procedure: Lumbar Puncture; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Procedure: Biopsy

INTERVENTIONS:
Biological: Odronextamab — Given IV
  Other Names: REGN1979; Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody REGN1979; WHO 11035
Procedure: Biospecimen Collection — Undergo collection of blood and oral or rectal swab samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Biological: Chimeric Antigen Receptor T-Cell Therapy — Undergo CAR-T cell therapy
  Other Names: CAR T Infusion; CAR T Therapy; CAR T-cell Therapy; Chimeric Antigen Receptor T-cell Infusion
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocyte Adsorptive Apheresis; Leukocytopheresis; Therapeutic Leukopheresis; White Blood Cell Reduction Apheresis
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: Bx

SUMMARY:
This phase II trial tests the effectiveness of odronextamab given before chimeric antigen receptor T (CAR-T) cell therapy (bridging therapy) in patients with large B-cell lymphomas that have come back after a period of improvement (relapsed) or that have not responded to previous treatment (refractory). Odronextamab is a bispecific antibody that can bind to two different antigens at the same time. Odronextamab binds to CD3, a T-cell surface antigen, and CD20 (a tumor-associated antigen that is expressed on B-cells during most stages of B-cell development and is often overexpressed in B-cell cancers) and may interfere with the ability of cancer cells to grow and spread. Bridging therapy has been used to maintain disease control and to increase the chance of successful receipt of CAR-T cell therapy. However, bridging therapy is typically given after leukapheresis, which does not help prevent disease progression between the decision for CAR-T cell therapy and leukapheresis. Giving odronextamab as bridging therapy before leukapheresis may delay disease progression to allow leukapheresis and increase the likelihood of successful CAR-T cell therapy in patients with relapsed or refractory large B-cell lymphomas.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive odronextamab intravenously (IV) on days 1, 2, 8, 9, 15 and 16 of cycle 1 (dose step-up), and on days 1, 8 and 15 of cycles 2-4 and then once every other week of remaining cycles. Cycles repeat every 21 days for the first 4 cycles, then every other week for up to a total of 12 months (including the first 2 cycles). After 2 cycles, patients undergo leukapheresis followed by lymphodepletion and CAR-T infusion per standard of care. If there is a significant delay of leukapheresis, patients may receive up to 12 additional weeks of treatment. Patients who achieve CR after cycle 2 may opt out of leukapheresis and CAR-T cell infusion and may continue to receive odronextamab in the absence of disease progression or unacceptable toxicity. Patients undergo positron emission tomography (PET)/computed tomography (CT), collection of blood and oral or rectal swab samples and tissue biopsy throughout the study. Additionally, patients may undergo lumbar puncture and bone marrow aspiration and/or biopsy on study.

After completion of study treatment, patients are followed till 90 days or the initiation of the next lymphoma directed therapy for toxicity check, and total duration of follow-up is up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed large B cell lymphoma, including diffuse large B-cell lymphoma (DLBCL) not otherwise specified, primary mediastinal large B-cell lymphoma, high grade B-cell lymphoma, DLBCL arising from indolent lymphoma, follicular lymphoma (FL) grade 3B
* Measurable disease, defined as at least one measurable lesion ≥ 15 mm on PET, CT, or magnetic resonance imaging (MRI) within one month of screening, according to the International Working Group consensus response evaluation criteria in lymphoma
* Prior frontline therapy for large B cell lymphoma must have failed the patient, and criteria must be met for receiving commercial axicabtagene ciloleucel (axi-cel), lisocabtagene maraleucel (liso-cel), or tisagenlecleucel (tisa-cel) per Food and Drug Administration (FDA) label
* Age ≥ 18 years
* Capable of understanding and providing a written informed consent
* Prior treatment with an anti-CD20 antibody therapy
* Eastern Cooperative Oncology Group performance status of 0-1; we allow enrollment of patients with a performance status of 2 if it is attributed to lymphoma per discretion of the treating physician or principal investigator (PI)
* Creatinine clearance ≥ 50 mL/min calculated by Cockcroft-Gault equation
* Total bilirubin ≤ 1.5 x the upper limit of normal (ULN), except in patients with Gilbert's syndrome
* Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x the ULN
* Adequate pulmonary function, defined as ≤ grade 1 dyspnea and oxygen saturation (SpO2) ≥ 92% on room air
* Adequate cardiac function, defined as left ventricular ejection fraction ≥ 50% and without evidence for pericardial effusion
* Platelet count ≥ 75 x 10^9 /L
* Hemoglobin (Hg) level ≥ 9 g/dL
* Absolute neutrophil count (ANC) ≥ 1 x 10^9 /L
* Patients with bone marrow involvement or splenic sequestration: Platelet count ≥ 25 x 10^9 /L
* Patients with bone marrow involvement or splenic sequestration: Hg ≥ 7.0 g/dL
* Patients with bone marrow involvement or splenic sequestration: ANC ≥ 0.5 x 10^9 /L
* Negative serum pregnancy test within 2 days of initiating odronextamab for women of childbearing potential (WOCBP), defined as those who have not been surgically sterilized or who have not been free of menses for at least 1 year
* Fertile male and WOCBP patients must be willing to use highly effective contraceptive methods from study recruitment to at least 6 months after the CAR T-cell infusion
* Patients must not provide egg or sperm donation until at least 6 months after the completion of the last dose of Odron

Exclusion Criteria:

* Detectable cerebrospinal fluid malignant cells, or brain metastases, or with a history of cerebrospinal fluid malignant cells or brain metastases
* History of a seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with central nervous system (CNS) involvement
* Standard anti-neoplastic chemotherapy (non-biologic) within 5-times the half-life or within 2 weeks, whichever is shorter, prior to first administration of study drug
* Standard radiotherapy within 2 weeks of first administration of study drug
* Prior treatment with an anti-CD20 x anti-CD3 bispecific therapy
* Allogeneic stem cell transplantation
* Any CAR-T cell therapy
* Patients may not be receiving other investigational agents
* Treatment with rituximab, alemtuzumab, or other investigational or commercial biologic agent within 2 weeks prior to first administration of study drug
* Immunosuppressive therapy (other than biologic) within 2 weeks of first administration of study drug
* Treatment with an investigational non-biologic agent within 2 weeks of first administration of study drug
* History of allergic reactions attributed to compounds of similar chemical or biologic composition of study drug
* History of hypersensitivity to any compound in the tetracycline antibiotics group
* Concurrent active malignancy for which the patient is receiving systemic treatment, unless approved by PI
* Known active and uncontrolled bacterial, viral, fungal, mycobacterial, or other infection
* Evidence of significant concurrent disease or medical condition that could interfere with the conduct of the study, or put the patient at significant risk including, but not limited to, significant cardiovascular disease (e.g., New York Heart Association class III or IV cardiac disease, myocardial infarction within the previous 6 months, unstable arrhythmias, or unstable angina) and/or significant pulmonary disease (e.g., obstructive pulmonary disease and history of symptomatic bronchospasm)
* Ongoing systemic corticosteroid treatment, with the exception of corticosteroid use for other (non-tumor and non-immunosuppressive) indications up to a maximum of 10 mg/day of prednisone or equivalent
* Infection with human immunodeficiency virus (unless viral load is undetectable and CD4 count ≥ 400) or chronic infection with hepatitis B virus or hepatitis C virus. Patients with hepatitis B (hepatitis B surface antigen positive [HepBsAg+]) with controlled infection were permitted upon consultation with the physician managing the infection
* Known hypersensitivity to both allopurinol and rasburicase
* Pregnant or breast-feeding women
* Administration of live vaccination within 28 days of first administration of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2028-04-10 (Estimated); Study Completion 2033-04-11 (Estimated)

PRIMARY OUTCOMES:
Failure to undergo leukapheresis | Up to 5 years
  Will include failures due to disease progression or adverse events (AEs) due to odronextamab (Odron), or requirement of other lymphoma-directed therapy for bridging before leukapheresis due to lack of response. Will report the total number and percentage with 95% confidence interval (CI).

SECONDARY OUTCOMES:
Receipt of chimeric antigen receptor T-cell therapy (CAR-T) | Up to 5 years
  Will estimate the total number and percentage with 95% CI of patients who receive CAR-T cell infusion. Patients who achieve complete response (CR) after 2 cycles of Odron and opt out of leukapheresis will be excluded from the estimation of the percentage. Will also report the reasons why patients do not eventually receive CAR-T.
Overall response rate (ORR) following bridging prior to CAR-T infusion | Up to 5 years
  ORR includes CR, partial response, stable disease. Will report the total number and percentage with 95% CI of patients who achieve response on positron emission tomography/computed tomography (PET/CT) scans before CAR-T cell infusion. Patients who receive CAR-T cell infusion will be included in the estimation of this percentage.
Progression free survival (PFS) following CAR-T infusion | Up to 2 years
  Will estimate the median with interquartile range of the progression free duration. Will also report the percentage with 95% CI.
CR rate | At 1 month after CAR-T
  Will report the total number and percentage with 95% CI of patients who achieve CR on the PET/CT scans following CAR-T cell infusion.
PFS in patients who achieve CR after 2 cycles of Odron, choose to opt out of CART, and receive up to a total of 12 months of Odron | Up to 5 years
  Will report the median duration of PFS with 95% CI in this group of patients.
Incidence of AEs | Up to 90 days after the last dose of Odron or the initiation of the next lymphoma directed therapy, whichever occurs first
  All AEs will be graded in severity according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0. Cytokine release syndrome and immune effector cell associated neurotoxicity syndrome will be graded by the American Society for Transplantation and Cellular Therapy Consensus Grading systems. Will report the rate and grade of each AE, including unsuccessful CAR-T production.

CONTACTS AND LOCATIONS:
Overall Officials: Mengyang Di, MD, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No